CLINICAL TRIAL: NCT06763120
Title: Prevelance and Risk Predictors of Post-operative Atrial Fibrillation Among Patients Undergoing Cardiac Surgery At Assiut University Heart Hospital
Brief Title: Post Operative Atrial Fibrillation Post Cardiac Surgery ( CABG and VALVE REPLACEMENT )
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa Allaam Moris Hakeem, Resident doctor, Assiut University
Other Study IDs: Post operative AF
Record Dates: First submitted 2024-12-15; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Atrial Fibrillation
Keywords: Post operative atrial fibrillation; Cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- First group is patients who developed post operative atrial fibrillation: Patients who developed post operative atrial fibrillation post CABG or valve replacement
- Second group is patients who don't develop post operative atrial fibrillation: Patient who don't develop post operative atrial fibrillation post CABG or valve replacement

SUMMARY:
This study aims to assess the percent and risk factors of postoperative atrial fibrillation in patients undergoing cardiac surgery in Assiut university heart hospital

DETAILED DESCRIPTION:
Arrhythmias are common complications after cardiac surgery, with postoperative atrial fibrillation (POAF) being the most frequently observed arrhythmia. The incidence rate of POAF ranges from 20% to 50%, depending on factors such as the type of surgery, patient population, and criteria used for diagnosis. Notably, POAF has been associated with increased morbidity, mortality, and health care costs. Patients who develop POAF are at a higher risk of experiencing complications such as stroke, heart failure (HF), and prolonged hospital stays. Moreover, POAF has been linked to long-term adverse outcomes, including a greater risk of recurrence of AF/atrial flutter and increased mortality. The accurate prediction of POAF can help guide therapy and facilitate targeted interventions to prevent its occurrence. Early identification of patients at risk for POAF allows for the timely initiation of prophylactic measures, such as the use of β-blockers, amiodarone, or other antiarrhythmic drugs, which have been shown to reduce the incidence of POAF. In this study we are searching for the percent and risk factors of POAF in patients undergoing cardiac surgery in Assiut university hospital.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years scheduled for first-time planned cardiac surgery ( CABG and Valve replacement)
2. Patients who are in sinus rhythm and not taking any antiarrhythmic medication, other than beta-adrenergic blocking agents, at the time of surgery.
3. Willingness to participate and provision of informed consent

Exclusion Criteria:

1. Prior history of cardiac surgery.
2. Pediatric population less than 18 years.
3. Patients with history of hyperthyroidism
4. Patients with electrolyte disturbance
5. Where follow-up is not possible.
6. The patient refused to sign the informed consent to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. ≥18 years scheduled for first-time planned cardiac surgery ( CABG and Valve replacement)
  2. Patients who are in sinus rhythm and not taking any antiarrhythmic medication, other than beta-adrenergic blocking agents, at the time of surgery.
  3. Willingness to participate and provision of informed consent
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Post operative atrial fibrillation | One year
  Prevelance of post operative atrial fibrillation in patients undergoing cardiac surgery ( past CABG and valve replacement )

CONTACTS AND LOCATIONS:
Overall Officials: Amr Ah Youssef, M,D, Study Chair — Assiut university heart hospital
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaPar DJ, Speir AM, Crosby IK, Fonner E Jr, Brown M, Rich JB, Quader M, Kern JA, Kron IL, Ailawadi G; Investigators for the Virginia Cardiac Surgery Quality Initiative. Postoperative atrial fibrillation significantly increases mortality, hospital readmission, and hospital costs. Ann Thorac Surg. 2014 Aug;98(2):527-33; discussion 533. doi: 10.1016/j.athoracsur.2014.03.039. PMID 25087786
- [Background] Villareal RP, Hariharan R, Liu BC, Kar B, Lee VV, Elayda M, Lopez JA, Rasekh A, Wilson JM, Massumi A. Postoperative atrial fibrillation and mortality after coronary artery bypass surgery. J Am Coll Cardiol. 2004 Mar 3;43(5):742-8. doi: 10.1016/j.jacc.2003.11.023. PMID 14998610
- [Background] Mathew JP, Fontes ML, Tudor IC, Ramsay J, Duke P, Mazer CD, Barash PG, Hsu PH, Mangano DT; Investigators of the Ischemia Research and Education Foundation; Multicenter Study of Perioperative Ischemia Research Group. A multicenter risk index for atrial fibrillation after cardiac surgery. JAMA. 2004 Apr 14;291(14):1720-9. doi: 10.1001/jama.291.14.1720. PMID 15082699
- [Background] Melduni RM, Schaff HV, Bailey KR, Cha SS, Ammash NM, Seward JB, Gersh BJ. Implications of new-onset atrial fibrillation after cardiac surgery on long-term prognosis: a community-based study. Am Heart J. 2015 Oct;170(4):659-68. doi: 10.1016/j.ahj.2015.06.015. Epub 2015 Jun 28. PMID 26386789